CLINICAL TRIAL: NCT03268408
Title: Impact Evaluation of the "Baby Newsletter" Project: an Intervention to Improve Parenting Self-efficacy in the First Year of Newborn's Life
Brief Title: Impact Evaluation of the "Baby Newsletter"
Acronym: BabyNewsletter
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: BabyNewsletter
Record Dates: First submitted 2017-08-23; First posted 2017-08-31 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2017-08

CONDITIONS: Parenting
Keywords: community intervention; newsletter

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intervention: Intervention aimed at improving self-efficacy parenting which consists in sending to new parents, during the first year of life of their son, eight newsletters with advices and recommendations on child care and development (project "Baby Newsletter").
  Interventions: Behavioral: Baby Newsletter
- Control: Usual care

INTERVENTIONS:
Behavioral: Baby Newsletter — eight newsletters sent home to newborns' parents with advices and recommendations on child care and development
  Groups: Intervention

SUMMARY:
Not-randomized controlled study to evaluate a community intervention to promote self-efficacy parenting. The treated group will be composed by all newborns resident in S.Ilario d'Enza (105 in 2013) where the Baby Newsletter is implemented. Newborns resident in the Health District of Montecchio and born in Montecchio Hospital in the same period are the control group (278 in 2013). Preterm or hospitalized children are excluded.

Self-efficacy parenting is evaluated through a questionnaire administered at baseline, after 5 and 12 months.

DETAILED DESCRIPTION:
Background

The importance of promoting parenting skills is worldwide recognized and, in Italy, different projects are implemented in order to develop these competences. The impact of these experiences is rarely evaluated.

The aim of this study is to evaluate the improvement in self-efficacy parenting produced by an intervention which consists in sending to every new parents, during the first year of life of their son, eight newsletters with advices and recommendations on child care and development (project "Baby Newsletter").

Methods

Not-randomized controlled study to evaluate a community intervention to promote self-efficacy parenting. The treated group will be composed by all newborns resident in S.Ilario d'Enza (105 in 2013) where the Baby Newsletter is implemented. Newborns resident in the Health District of Montecchio and born in Montecchio Hospital in the same period are the control group (278 in 2013). Preterm or hospitalized children are excluded.

Self-efficacy parenting is evaluated through the TOPSE (Tool to measure Parenting Self-Efficacy) questionnaire administered at baseline, in Montecchio Birth Unit or at the paediatric clinics, and at the vaccination appointments after 5 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* being parent of a child born during the study enrollment period and resident in the Montecchio Health District
* good comprehension of Italian language

Exclusion Criteria:

* delivering in other facilities than the Montecchio hospitals (only for controls)
* parents of newborns with pathological conditions at born
* parents of newborns that were transferred to another hospital immediately after born due to clinical reasons
* parents of pre-term newborns

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: * Newsletter Group
    * all the parents of newborns delivered during the study period (01/09/2014 - 31/12/2015) resiident in the Sant'Ilario municipality.
  * Control Group
    * all the parents f newborns delivered during the study period (01/09/2014 - 31/12/2015) resident in other municipalities of the Montecchio health district
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Parenting score on the scale "emotion and affection" | 12 months
  score based on 6 items of TOPSE questionnaire
Parenting score on the scale "play and enjoyment" | 12 months
  score based on 6 items of TOPSE questionnaire
Parenting score on the scale "empathy and understanding" | 12 months
  score based on 6 items of TOPSE questionnaire
Parenting score control | 12 months
  score based on 6 items of TOPSE questionnaire
Parenting score on the scale "discipline and setting boundaries" | 12 months
  score based on 6 items of TOPSE questionnaire
Parenting score pressures | 12 months
  score based on 6 items of TOPSE questionnaire
Parenting score self-acceptance | 12 months
  score based on 6 items of TOPSE questionnaire
Parenting score on the scale "learning and knowledge" | 12 months
  score based on 6 items of TOPSE questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Costantino Panza, MD, Principal Investigator — AUSL Reggio Emilia
Locations (1):
- Montecchio Hospital, Montecchio Emilia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kendall S, Bloomfield L. Developing and validating a tool to measure parenting self-efficacy. J Adv Nurs. 2005 Jul;51(2):174-81. doi: 10.1111/j.1365-2648.2005.03479.x. PMID 15963189
- [Derived] Panza C, Volta A, Broccoli S, Bonvicini L, Kendall S, Marchesi M, Giorgi Rossi P. Evaluation of an intervention aimed at supporting new parents: the Baby Newsletter project. Ital J Pediatr. 2020 Sep 4;46(1):123. doi: 10.1186/s13052-020-00886-5. PMID 32887637